CLINICAL TRIAL: NCT03230318
Title: A Pivotal Study of Derazantinib in Patients With Inoperable or Advanced Intrahepatic Cholangiocarcinoma and FGFR2 Gene Fusions or FGFR2 Gene Mutations or Amplifications
Brief Title: Derazantinib in Subjects With FGFR2 Gene Fusion-, Mutation- or Amplification- Positive Inoperable or Advanced Intrahepatic Cholangiocarcinoma
Acronym: FIDES-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZB-CS-301; ARQ 087-301 (Other: ArQule, Inc)
Expanded Access: NCT04087876 (No longer available)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Intrahepatic Cholangiocarcinoma; Combined Hepatocellular and Cholangiocarcinoma
Keywords: iCCA; intrahepatic cholangiocarcinoma; FGFR2 gene fusion or FGFR2 gene mutation or amplification; biliary cancer; bile duct cancer; FGFR2 gene rearrangement; liver cancer; targeted therapy; combined hepatocellular and cholangiocarcinoma; cHCC-CCA; derazantinib
MeSH Terms: conditions — Cholangiocarcinoma; Liver Neoplasms; Biliary Tract Neoplasms; Bile Duct Neoplasms | interventions — derazantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- derazantinib (Experimental): Oral administration
  Interventions: Drug: derazantinib

INTERVENTIONS:
Drug: derazantinib — Derazantinib was administered orally at 300 mg once daily

SUMMARY:
This Phase II, open-label, single-arm study evaluated the anti-cancer activity of derazantinib in subjects with inoperable or advanced intrahepatic cholangiocarcinoma (iCCA) who received at least one prior regimen of systemic therapy. Patients received an oral once-daily total dose of 300 mg derazantinib capsules.

DETAILED DESCRIPTION:
This was a multi-center, open-label, single arm study which evaluated the anti-cancer activity of derazantinib in adult patients with inoperable or advanced iCCA in the following study population:

Patients with inoperable or advanced iCCA and with fibroblast growth factor receptor 2 (FGFR2) fusions (Substudy 1) or FGFR2 mutations/amplifications (Substudy 2), treated with at least one prior regimen of systemic therapy.

Derazantinib was supplied as 100 mg capsules. A dose of 300 mg once-daily (three capsules of 100 mg each) of derazantinib was administered orally to patients, 1 hour before, or 2 hours after, a meal.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed written informed consent granted prior to initiation of any study-specific procedures
2. 18 years of age or older
3. Histologically or cytologically confirmed locally advanced, inoperable, or metastatic iCCA or mixed histology tumors
4. Substudy 1:

   FGFR2 fusion status based on the following assessments:

   a) If central laboratory was designated by Sponsor: Positive FISH test; and/or b) If non-central laboratory: i) Positive FISH or NGS test: patients were potentially enrolled and started dosing, but central confirmation was required* ii) Negative FISH or NGS test: tissue was submitted to the central laboratory designated by the Sponsor, and patients were only enrolled in case the central test was positive

   *By used standard protocols and approved by local IRB/EC, by CLIA or other similar agency.

   Substudy 2:

   FGFR2 mutation/amplification status based on local NGS testing performed or commissioned by the respective study site.
5. Received at least one regimen of prior systemic therapy and then experienced documented radiographic progression
6. Measurable disease by RECIST version 1.1 criteria
7. ECOG performance status ≤ 1
8. Adequate organ functions as indicated by the following laboratory values (based on screening visit values from the central laboratory).

   * Hematological

     * Hemoglobin (Hgb) ≥ 9.0 g/dL
     * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
     * Platelet count ≥ 75 x 109/L
     * International normalized ratio (INR) 0.8 to upper limit of normal (ULN) or ≤ 3 for subjects who received anticoagulant therapy such as Coumadin or heparin
   * Hepatic

     * Total bilirubin ≤ 2 x ULN
     * AST and ALT ≤ 3 ULN (≤ 5 x ULN for subjects with liver metastases)
     * Albumin ≥ 2.8 g/dL
   * Renal

     * Serum creatinine ≤ 1.5 x ULN
     * Creatinine clearance of ≥ 30 mL/min as estimated by the Cockcroft-Gault equation
9. Female and male patients of child-producing potential must had agreed to avoid becoming pregnant or impregnating a partner, respectively, used double-barrier contraceptive measures, oral contraception, or had to avoid of intercourse, during the study, and until at least 120 for 90 days after the last dose of derazantinib.

Male or female patients of child-producing potential must had agreed to comply with one of the following until at least 120 days after the last dose of derazantinib:

1. Abstinence from heterosexual activity
2. Using (or having their partner use) an acceptable method of contraception during heterosexual activity.

Key Exclusion Criteria:

1. Receipt of treatment before the first dose of study drug (Cycle 1 Day 1) within an interval shorter than the following, as applicable:

   * One chemotherapy or biological (e.g., antibody) cycle interval
   * Five half-lives of any small-molecule investigational or licensed medicinal product
   * Two weeks, for any investigational medicinal product with an unknown half-life
   * Four weeks of curative radiotherapy
   * Seven days of palliative radiotherapy
   * 28 days of radiotherapy
2. Major surgery, locoregional therapy, or radiation therapy within four weeks of the first dose of derazantinib
3. Previous treatment with any FGFR inhibitor (e.g., Balversa® [erdafitinib], Pemazyre® [pemigatinib], infigratinib, rogaratinib, futibatinib, lenvatinib, ponatinib, dovitinib, nintedanib, AZD4547, LY2784455).
4. Patients who were unable or unwilling to swallow the complete daily dose of derazantinib capsules
5. Clinically unstable central nervous system (CNS) metastases (to be eligible, subjects must had stable disease ≥ 3 months, confirmed by magnetic resonance imaging (MRI) or computed tomography (CT) scan, and/or had CNS metastases well controlled by low-dose steroids, anti-epileptics, or other symptom-relieving medications)
6. Evidence of clinically significant corneal or retinal disorder which was likely to increase the risk of eye toxicity, including but not limited to bullous/band keratopathy, keratoconjunctivitis (unless keratoconjunctivitis sicca), corneal abrasion, inflammation/ulceration, confirmed by ophthalmologic examination.
7. Uncontrolled or active hepatobiliary disorders, untreated or ongoing complications after laparoscopic procedures or stent placement, including but not limited to active cholangitis, biloma or abscess (to be eligible, the subjects had to be treated and disorders/complications should had been resolved within 2 weeks prior to the first dose of derazantinib)
8. History of significant cardiac disorders:

   * Myocardial infarction (MI) or congestive heart failure defined as Class II to IV per the New York Heart Association (NYHA) classification within 6 months of the first dose of derazantinib (MI that occurred > 6 months prior to the first dose of derazantinib was permitted)
   * QTcF >450 msec (males or females)
9. Serum electrolyte abnormalities defined as follows:

   * Hyperphosphataemia: Serum phosphate > institutional ULN
   * Hyperkalemia: > 6.0 mmol/L
   * Hypokalemia: < 3.0 mmol/L
   * Hypercalcemia: corrected serum calcium < 1.75 mmol/L (< 7.0 mg/dL)
   * Hypocalcemia: corrected serum calcium > 3.1 mmol/L (> 12.5 mg/dL)
   * Hypomagnesemia: < 0.4 mmol/L (< 0.9 mg/dL)
10. Significant gastrointestinal disorder(s) that could had, in the opinion of the Investigator, interfered with the absorption, metabolism, or excretion of derazantinib (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection)
11. History of additional malignancy that was progressing or required active treatment. Exceptions included basal cell carcinoma of the skin, squamous cell carcinoma of the skin that had undergone potentially curative therapy, and in situ cervical cancer.
12. Uncontrolled illness not related to cancer, including but not limited to:

    * Psychiatric illness/substance abuse/social situation that would limit compliance with study requirements
    * Known uncontrolled human immunodeficiency virus (HIV) infection
    * Severe bacterial, fungal, viral and/or parasitic infections on therapeutic oral or IV medication at the time of first dose of study drug administration
13. Blood or albumin transfusion within 5 days of the blood draw which has been used to confirm eligibility
14. Pregnant or breast feeding
15. Known hypsersensitivity to derazantinib, or to any of the study drug excipients (starch, lactose, crospovidone, magnesium stearate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Häckl, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (41):
- United States (11):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center - Sidney Kimmel Center for Prostate and Urologic Cancers, New York, New York
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
- Belgium (3):
  - Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
- France (2):
  - CHU Grenoble Alpes, La Tronche
  - Gustave Roussy, Villejuif
- Germany (5):
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- St. James's Hospital, Dublin, Ireland
- Italy (6):
  - Sant'Orsola-Malpighi Hospital, University of Bologna, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale San Gerardo, Monza
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Humanitas Cancer Center, Istituto Clinico Humanitas IRCCS, Rozzano
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (4):
  - Vall d'Hebrón University Hospital, Barcelona
  - Catalan Institute of Oncology, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Universitätsspital Basel, Basel, Switzerland
- United Kingdom (3):
  - University College London Hospitals NHS Foundation Trust, Euston
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Marsden, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazzaferro V, El-Rayes BF, Droz Dit Busset M, Cotsoglou C, Harris WP, Damjanov N, Masi G, Rimassa L, Personeni N, Braiteh F, Zagonel V, Papadopoulos KP, Hall T, Wang Y, Schwartz B, Kazakin J, Bhoori S, de Braud F, Shaib WL. Derazantinib (ARQ 087) in advanced or inoperable FGFR2 gene fusion-positive intrahepatic cholangiocarcinoma. Br J Cancer. 2019 Jan;120(2):165-171. doi: 10.1038/s41416-018-0334-0. Epub 2018 Nov 13. PMID 30420614

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 729 patients underwent molecular screening, and 148 were enrolled and assigned treatment. One patient was subsequently not confirmed to have fibroblast growth factor receptor 2 (FGFR2) fusion, and was therefore excluded from the Safety/ITT population, meaning that for all Safety/ITT population analyses 147 patients were included (Substudy 1 = 103, Substudy 2 = 44).
Groups:
- Substudy 1: Substudy 1 comprised of patients with inoperable or advanced iCCA with FGFR2 fusions
  Derazantinib was administered orally at 300 mg once daily
- Substudy 2: Substudy 2 comprised of patients with with inoperable or advanced iCCA with FGFR2 mutations or amplifications
  Derazantinib was administered orally at 300 mg once daily
Period: Overall Study
Arm/Group | Substudy 1 | Substudy 2
Started | 104 | 44
Completed | 0 | 0
Not Completed | 104 | 44
Not completed — Radiographic disease progression | 72 | 19
Not completed — Clinical progression | 17 | 7
Not completed — Adverse Event | 5 | 3
Not completed — Physician Decision | 2 | 3
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Other | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Substudy 2: Substudy 2 comprised of patients with inoperable or advanced iCCA with FGFR2 mutations or amplifications
  Derazantinib was administered orally at 300 mg once daily
- Total: Total of all reporting groups
Arm/Group | Substudy 1 | Substudy 2 | Total
Number analyzed (Participants) | 103 | 44 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.28) | 61.3 (11.75) | 58.0 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 25 | 92
  Male | 36 | 19 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 0 | 8
  White | 86 | 37 | 123
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Substudy 1: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of patients who achieved a confirmed clinical response (CR) or partial response (PR) by blinded independent central review using the internationally recognized criteria for the radiological assessment in tumor response of solid tumors (RECIST) Version 1.1
Time Frame: From first dose and up to 54 months
Population: Intent-to-treat (ITT) Population: included all patients who received any amount of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy 1
Number analyzed (Participants) | 103
Percentage of participants | 22.3 [14.7 to 31.6]

2. Primary Outcome: Substudy 2: Progression Free Survival at 3 Months (PFS 3)
Description: PFS3 was defined as the proportion of patients who have progression-free survival at 3 months from the first date of receiving study drug as assessed by survival status and blinded independent central review as per RECIST 1.1.
Time Frame: From first dose and up to 3 months
Population: Modified intent-to-treat (mITT) Population: included all patients in the Safety/ITT population, who had at least one post-baseline disease assessment (at least one post-baseline imaging assessment in accordance with RECIST 1.1, or documented clinical progression [every effort was made to objectively assess radiographic progression]), or reported death during the treatment period.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy 2
Number analyzed (Participants) | 43
Percentage of participants | 62.8 [46.7 to 77.0]

3. Secondary Outcome: PFS
Description: PFS was calculated from the first date of receiving study drug until radiographic disease progression by blinded independent central review or death.
Time Frame: From first dose and up to 54 months
Population: mITT Population: included all patients in the Safety/ITT population, who had at least one post-baseline disease assessment (at least one post-baseline imaging assessment in accordance with RECIST 1.1, or documented clinical progression [every effort was made to objectively assess radiographic progression]), or reported death during the treatment period.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Substudy 1: Substudy 1 comprised of patients with iCCA with FGFR2 fusions
  Derazantinib was administered orally at 300 mg once daily one hour prior to or two hours after a meal
- Substudy 2: Substudy 2 comprised of patients with iCCA with FGFR2 mutations or amplifications
  Derazantinib was administered orally at 300 mg once daily one hour prior to or two hours after a meal
Arm/Group | Substudy 1 | Substudy 2
Number analyzed (Participants) | 103 | 44
Months | 8.1 [5.5 to 8.3] | 8.3 [3.5 to NA] — Not evaluable due to the insufficient number of events

4. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated from the first date of receiving study drug until death
Time Frame: From first dose and up to 54 months
Population: ITT population: included all patients who received any amount of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Substudy 1 | Substudy 2
Number analyzed (Participants) | 103 | 44
Months | 17.2 [12.5 to 22.4] | 11.9 [8.4 to 15.9]

5. Secondary Outcome: Duration of Response (DoR)
Description: DoR was calculated from the first date of documented tumor response to disease progression by blinded independent central review per RECIST version 1.1 DoR was derived only for patients who have the best overall response of CR or PR
Time Frame: From first dose and up to 54 months
Population: ITT Population: included all patients who received any amount of study drug
Measure: Median (Full Range); unit: Months
Arm/Group | Substudy 1 | Substudy 2
Number analyzed (Participants) | 103 | 44
Months | 6.5 [4.6 to 9.2] | NA [NA to NA] — Not evaluable due to the insufficient number of events

6. Secondary Outcome: Substudy 2: Objective Response Rate
Description: as for outcome 1
Time Frame: From first dose and up to 54 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy 2
Number analyzed (Participants) | 43
Percentage of participants | 9.3 [2.6 to 22.1]

7. Secondary Outcome: Number of Patients With Grade 3-5 Treatment-emergent Adverse Events (TEAEs)
Description: Number of patients experiencing TEAE of Grade 3 to 5 according to Common Terminology Criteria for Adverse Events (CTCAE)
Time Frame: TEAEs were defined as all events occurring after drug treatment began and up to 30 days after last study drug administration
Population: Safety / ITT population included all patients who received any amount of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy 1 | Substudy 2
Number analyzed (Participants) | 103 | 44
Participants
  Number of patients with only unrelated TEAEs of Grade 3-5 | 31 | 16
  Number of patients with related TEAEs of Grade 3-5 | 35 | 10
  Number of patients without TEAEs of Grade 3-5 | 37 | 18

ADVERSE EVENTS:
Time Frame: All AEs were assessed from first day of treatment and until 28-35-day post-treatment follow-up period. The AE assessment period for the whole study lasted up to 50 months.
Arm/Group | Substudy 1 | Substudy 2
All-Cause Mortality (participants affected / at risk) | 74/103 | 25/44
Serious Adverse Events (participants affected / at risk) | 37/103 | 16/44
Other Adverse Events (participants affected / at risk) | 103/103 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substudy 1 (N=103) | Substudy 2 (N=44)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liver transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 9 (9) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Substudy 1 (N=103) | Substudy 2 (N=44)
Alanine aminotransferase increased (Investigations) | 36 (43) | 13 (15)
Aspartate aminotransferase increased (Investigations) | 46 (52) | 13 (15)
Blood alkaline phosphatase increased (Investigations) | 17 (18) | 9 (11)
Blood creatinine increased (Investigations) | 17 (18) | 7 (8)
Blood phosphorus increased (Investigations) | 13 (20) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (6) | 3 (3)
Platelet count decreased (Investigations) | 10 (20) | 5 (5)
Weight decreased (Investigations) | 17 (17) | 6 (6)
White blood cell count decreased (Investigations) | 6 (11) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 16 (18) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (8) | 1 (1)
Dizziness (Nervous system disorders) | 13 (13) | 3 (3)
Dysgeusia (Nervous system disorders) | 20 (20) | 11 (11)
Headache (Nervous system disorders) | 12 (14) | 5 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 8 (9) | 1 (1)
Cornea verticillata (Eye disorders) | 7 (7) | 1 (1)
Dry eye (Eye disorders) | 20 (20) | 7 (7)
Keratitis (Eye disorders) | 2 (2) | 3 (3)
Vision blurred (Eye disorders) | 26 (26) | 6 (8)
Visual acuity reduced (Eye disorders) | 7 (7) | 0 (0)
Visual impairment (Eye disorders) | 5 (5) | 3 (4)
Xerophthalmia (Eye disorders) | 9 (11) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 26 (30) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 10 (12) | 1 (1)
Constipation (Gastrointestinal disorders) | 28 (31) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 34 (52) | 14 (21)
Dry mouth (Gastrointestinal disorders) | 30 (32) | 17 (17)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 1 (2)
Nausea (Gastrointestinal disorders) | 41 (51) | 18 (23)
Vomiting (Gastrointestinal disorders) | 30 (43) | 15 (23)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (17) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (14) | 3 (3)
Nail discolouration (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 20 (23) | 9 (9)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 11 (11) | 3 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 30 (36) | 12 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (9) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (8) | 4 (4)
Vitamin D deficiency (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 9 (9) | 2 (3)
Hypertension (Vascular disorders) | 24 (30) | 5 (7)
Asthenia (General disorders) | 25 (27) | 6 (8)
Fatigue (General disorders) | 34 (37) | 13 (16)
Mucosal inflammation (General disorders) | 3 (3) | 3 (3)
Oedema peripheral (General disorders) | 5 (5) | 4 (5)
Pyrexia (General disorders) | 7 (9) | 2 (2)
Anxiety (Psychiatric disorders) | 8 (8) | 2 (2)
Depression (Psychiatric disorders) | 7 (7) | 1 (1)
Insomnia (Psychiatric disorders) | 15 (15) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT03230318/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/18/NCT03230318/SAP_001.pdf